CLINICAL TRIAL: NCT07356999
Title: Characterization of Visual Perception Alterations in Patients With Idiopathic Scoliosis: Towards a Theory of Perceptual Imbalance
Brief Title: Characterization of Visual Perception Impairments in Patients With Idiopathic Scoliosis
Acronym: EYAIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Médico-Chirurgical de Réadaptation des Massues Croix Rouge Française (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025_10_EYAIS_RIPH2; 2025-A01301-48 (Other: ANSM)
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Scoliosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vertical Perception Assessment (Experimental)
  Interventions: Other: Motion Analysis

INTERVENTIONS:
Other: Motion Analysis — Researchers use motion capture to track exactly how a patient's body moves and shifts in response to different environments.

SUMMARY:
Scoliosis is more than just a curve in the spine; it is a complex, 3D twisting of the backbone. While it can be caused by birth defects or tumors, the most common type-idiopathic scoliosis-appears in healthy teenagers for no clearly known reason.

The Theory of Balance Researchers believe that scoliosis might actually be caused by a "glitch" in how the body stays upright. Instead of the spine curving on its own, the curve might be the body's way of compensating for a poor sense of balance.

To stay balanced, the human brain relies on three main "inputs":

1. The Vestibular System: Located in the inner ear (detects movement).
2. Proprioception: The body's "inner map" (sensing where your limbs are).
3. Vision: Seeing the world around you to stay oriented.

The Goal of the Study Even though humans rely heavily on their eyes to stay balanced, the role of vision in scoliosis has not been studied very much.

This experiment aims to test the hypothesis that teenagers with scoliosis have trouble processing visual information to maintain their posture. By using advanced motion analysis, researchers want to see if a "misunderstanding" of visual cues is contributing to the spinal deformity.

ELIGIBILITY:
Inclusion Criteria:

Group Scoliosis:

* Girls or boys aged 11 to 18 inclusive.
* Patients with progressive idiopathic scoliosis
* Candidates for either orthopedic (brace) or surgical (arthrodesis correction) treatment for which a pre-therapeutic multimodal assessment is planned.

Control group:

- Girls or boys aged 11 to 18 inclusive.

Exclusion Criteria:

The following individuals will not be included:

* Individuals with another musculoskeletal disorder.
* Individuals with a neurosensory disorder that may affect the balance of the trunk or lower limbs.
* Individuals with uncorrected visual perception disorders (visual check within 12 months prior to the examination).
* Lack of consent from the subject.
* Lack of consent from legal representatives.
* Failure to understand the instructions for performing the tests.

In addition, for the control group:

- Suffering from scoliosis

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Margin of Dynamic Stability | At enrollment
  This measures how close a person is to losing their balance while moving. It calculates the distance between where the body's weight is moving and the edge of the person's "footprint" (base of support).
Center of Pressure | At enrollment
  The point on the ground where the most weight is being concentrated. Tracking how much this point "wobbles" or shifts shows how hard the body is working to stay upright.
Extrapolated Center of Mass | At enrollment
  A calculation that looks at both the position of the body and its velocity. It helps researchers predict if the person's momentum is about to carry them off-balance.

SECONDARY OUTCOMES:
Base of Support | At enrollment
  The total area on the ground occupied by the feet. A wider BoS often suggests the subject is trying to create a "wider stance" to feel more stable.
Visual Field Perception | At enrollment
  The "Distance Error." Using a joystick, the patient tries to place a 3D avatar exactly halfway between two other figures. The difference between the true middle and where the patient thinks the middle is reveals if their depth perception is distorted.
Subjective Visual Vertical | At enrollment
  Angular Error. A glowing line is tilted on a screen, and the patient must tell the operator how to rotate it until it is perfectly vertical.